CLINICAL TRIAL: NCT00000687
Title: Phase II Study of Zidovudine and Recombinant Alpha-2A Interferon in the Treatment of Patients With AIDS-Associated Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 096; 11071 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Interferon Alfa-2a; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Interferon alpha-2; Zidovudine

INTERVENTIONS:
Drug: Interferon alfa-2a
Drug: Zidovudine

SUMMARY:
To determine the safety and effectiveness of combining zidovudine (AZT) and interferon alfa-2a (IFN-A2a) in a treatment for Kaposi's sarcoma (KS) in patients who have AIDS. It is hoped with the present study to define the rate at which the treatment affects the tumors and also to assess any toxic effects of the combination treatment over a period of time.

In a recent study, the combination of IFN-A2a and AZT in the treatment of patients with AIDS-associated KS was evaluated and safe doses of both AZT and IFN-A2a were determined. In addition, it appeared that there was a substantial reduction in KS lesions with this therapy. Potential benefits of this combined therapy include resolution of KS lesions, prolonged survival, a decrease in the frequency and severity of opportunistic infections, improvement in CD4 cells, and a decrease in serum p24 antigens.

DETAILED DESCRIPTION:
In a recent study, the combination of IFN-A2a and AZT in the treatment of patients with AIDS-associated KS was evaluated and safe doses of both AZT and IFN-A2a were determined. In addition, it appeared that there was a substantial reduction in KS lesions with this therapy. Potential benefits of this combined therapy include resolution of KS lesions, prolonged survival, a decrease in the frequency and severity of opportunistic infections, improvement in CD4 cells, and a decrease in serum p24 antigens.

Following evaluation studies, patients who participate in the study receive IFN-A2a and AZT. IFN-A2a is administered as a single subcutaneous injection once a day. AZT is given in a single capsule every 4 hours through the day for a total of six capsules. The first phase of treatment continues for 8 weeks followed by a 1-week rest period, during which time AZT only is given. Subjects who have had an interruption in interferon during the first 8 weeks of the study for a toxicity may skip the rest period. Patients experiencing a complete response will be placed on maintenance therapy. Patients without progression of their KS can continue on the treatment of AZT and IFN-A2a until a complete response is obtained or until study is terminated, whichever comes first. Patients with complete anti-tumor response can continue on a maintenance phase, in which they receive IFN-A2a as a single injection 3 times a week on nonconsecutive days and a single capsule of AZT q4h 6 x /day until the study is terminated on February 1, 1992. Patients are required to visit the clinic weekly for the first 12 weeks (except during the week 9 rest period), every other week for the next 8 weeks, every month for up to 52 weeks of the study and every 3 months thereafter. Throughout the study, frequent blood samples will be taken to monitor the effectiveness and safety of the treatment.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Inhalation pentamidine for the prevention of Pneumocystis carinii pneumonia (PCP) at a dose of 300 mg once every 4 weeks.
* AMENDED: Trimethoprim - sulfamethoxazole or dapsone only if on the maintenance phase of the study.

Concurrent Treatment:

Allowed:

* Blood transfusions.

Patients must have a positive antibody to HIV by any federally licensed ELISA test. All lab tests must be within 7 days of entry into the study.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Other antiretroviral agents.
* Immunomodulators.
* Corticosteroids.
* Cytotoxic chemotherapy.
* Aspirin.
* H2 blockers.
* Barbiturates and myelosuppressive drugs should be particularly avoided as they may interfere with the metabolism or enhance the toxicities of either zidovudine or interferon alfa-2a.
* Other experimental medications.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with prior experience of Grade 4 toxicity to zidovudine therapy will be excluded from the study.

Prior Medication:

Excluded:

* Interferon therapy.
* Excluded within 30 days of study entry:
* Immunomodulators.
* Corticosteroids.
* Cytotoxic chemotherapeutic agents.
* Excluded within 14 days of study entry:
* Zidovudine (AZT).

Prior Treatment:

Excluded within 30 days of study entry:

* Blood transfusions.
* Radiation therapy.

Patients may not have any of the following diseases or symptoms:

* Active opportunistic infection associated with AIDS.
* Significant neurologic disease associated with AIDS, as manifested by motor abnormalities including impaired rapid eye movement or ataxia, motor weakness in the lower extremities, sensory deficit consistent with a peripheral neuropathy, bladder or bowel incontinence.
* Internal organ involvement with Kaposi's sarcoma, i.e., nonnodal visceral Kaposi's sarcoma, excluding minimal gastrointestinal disease of less than 5 lesions.
* Tumor-associated edema.
* Current neoplasm other than Kaposi's sarcoma.
* Significant cardiac disease, including a recent history of myocardial infarction or significant current cardiac arrhythmias.

Active drug or alcohol abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Study Completion 1993-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Fischl, Study Chair
Locations (9):
- United States (9):
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Fischl MA, Finkelstein DM, He W, Powderly WG, Triozzi PL, Steigbigel RT. A phase II study of recombinant human interferon-alpha 2a and zidovudine in patients with AIDS-related Kaposi's sarcoma. AIDS Clinical Trials Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Apr 1;11(4):379-84. doi: 10.1097/00042560-199604010-00008. PMID 8601224